CLINICAL TRIAL: NCT00573885
Title: Phase II Trial of Polyphenon E in Former Smokers With Abnormal Sputa
Brief Title: Green Tea Extract in Preventing Cancer in Former and Current Heavy Smokers With Abnormal Sputum
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000578191; P01CA096964 (NIH); BCCA-H03-61083; BCCA-R03-1083
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Tobacco Use Disorder
Keywords: non-small cell lung cancer; small cell lung cancer; tobacco use disorder
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral defined green tea catechin extract twice daily for 6 months.
  Interventions: Drug: defined green tea catechin extract
- Arm II (Placebo Comparator): Patients receive oral placebo twice daily for 6 months.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: defined green tea catechin extract — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. Green tea extract may keep cancer from forming.

PURPOSE: This randomized phase II trial is studying green tea extract in preventing cancer in former and current heavy smokers with abnormal sputum.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy and safety of defined green tea catechin extract (polyphenon E) in former smokers with abnormal sputum score using stringent, newly developed response criteria of combined nuclear morphometry and malignancy-associated changes as the primary surrogate endpoint.
* Evaluate if polyphenon E can modulate other surrogate endpoint biomarkers of aberrant methylation, cell cycle regulation, apoptosis, oncogene/tumor suppressor gene expression, as well as phase I and II enzyme regulation.
* Establish a library of in-vivo confocal micro-endoscopy and optical coherent tomography images of the bronchial epithelium with corresponding histopathology, nuclear morphometry, and other biomarker information to assess the potential of confocal micro-endoscopy as a non-biopsy method to assess the effect of chemoprevention agents.

OUTLINE: This is an open label, part 1 study followed by a randomized, double-blind, part 2 study.

* Part 1 (completed March 22, 2006): Patients receive oral defined green tea catechin extract twice daily in months 1 and 2 and inhaled budesonide twice daily in month 2.

Patients undergo autofluorescence bronchoscopy with biopsies, oral and bronchial brushing, and bronchoalveolar lavage at the end of months 1 and 2.

* Part 2: Patients are stratified by gender and randomized to 1 of 2 treatment arms.

  * Arm I: Patients receive oral defined green tea catechin extract twice daily for 6 months.
  * Arm II: Patients receive oral placebo twice daily for 6 months. Patients who have progressive or stable disease at 6 months may receive open-label defined green tea catechin extract.

Patients undergo autofluorescence bronchoscopy with biopsies, oral and bronchial brushing, and bronchoalveolar lavage at the end of months 6 and 12.

Blood samples are collected periodically for biomarker studies. After completion of study therapy, patients are followed periodically for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Current smokers who have smoked at least 30 pack-years (e.g., 1 pack per day for 30 years or more) (part 1; completed March 22, 2006)
* Former smokers who have smoked at least 30 pack-years (part 2)

  * A former smoker is defined as one who has stopped smoking for one or more years
* Abnormal sputum score ≥ 0.25 by computer-assisted image analysis
* Exhaled carbon monoxide level < 5 ppm (part 2 )
* Willing to take defined green tea catechin extract/placebo twice a day regularly
* No evidence of overt lung cancer

  * No carcinoma in situ or invasive cancer on bronchoscopy or abnormal spiral chest CT suspicious of lung cancer

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine normal
* Bilirubin normal
* AST and ALT normal
* Alkaline phosphatase normal

Exclusion criteria:

* Chronic active hepatitis/liver cirrhosis
* Severe heart disease (e.g., unstable angina, chronic congestive heart failure, use of antiarrhythmic agents)
* Ongoing gastric ulcer
* Acute bronchitis or pneumonia within one month
* Known reaction to lidocaine, albuterol sulfate, midazolam hydrochloride, and/or alfentanil hydrochloride
* Known allergy to green tea and/or corn starch, gelatin, or other nonmedicinal ingredients
* Any medical condition, such as acute or chronic respiratory failure or bleeding disorder that, in the opinion of the investigator, could jeopardize the patient's safety during participation in the study
* Unwilling to have a bronchoscopy
* Unwilling to have a spiral chest CT

PRIOR CONCURRENT THERAPY:

* No more than 5 cups of tea a week
* No concurrent anticoagulant treatment such as warfarin or heparin
* No use of other natural health products containing green tea compounds

Ages: 45 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Changes in oncogene/tumor suppression gene expression (part 1; completed March 22, 2006) | 36 months
Phase I and II enzyme regulation by Affymetrix chip analysis in bronchial brush cells (part 1) | 60 months
C-reactive protein level in plasma before treatment and 1 and 2 months after treatment (part 1) | 60 months
Quantitative sputum score by image analysis before and 6 months after treatment (part 2) | 36 months

SECONDARY OUTCOMES:
Change in pathology grade of bronchial biopsies (part 2) | 36 months
Morphometric index of bronchial biopsies and bronchoalveolar lavage cells (BAL) (part 2) | 36 months
Methylation markers in sputa and BAL cells (part 2) | 60 months
Ki-67 expression (part 2) | 60 months
Cleaved caspase 3, p53, and VEGF assays in bronchial biopsies (part 2) | 60 months
Oncogene and tumor suppression gene expression (part 2) | 60 months
Phase I and II enzyme regulation by Affymetrix chip analysis of RNA from bronchial brush cells (part 2) | 60 months
C-reactive protein levels in plasma before treatment, and 6 months after treatment (part 2) | 36 months
Resolution or progression of non-calcified lung nodules on spiral CT (part 2) | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Lam, MD, Study Chair — British Columbia Cancer Agency
Locations (1):
- British Columbia Cancer Agency - Vancouver Cancer Centre, Vancouver, British Columbia, Canada